CLINICAL TRIAL: NCT04658069
Title: T Cell Dysfunction in End-stage Renal Disease
Brief Title: T Cell Dysfunction in ESRD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TcdiESRD
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: ESRD; T-Cell Dysfunction
Keywords: T cell dysfunction; end-stage renal disease; clinical outcome
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One Cohort receiving routine hemodialysis therapy without any specific interventions: all HD patients enrolled in this study
  Interventions: Other: no specific interventions

INTERVENTIONS:
Other: no specific interventions — no specific interventions

SUMMARY:
Patients with end-stage renal disease (ESRD) suffer from high morbidity and mortality of cardiovascular and infectious disease and increased risk of all-cause mortality which is mainly attributed to the disturbed immune response. More and more evident indicated that T cell dysfunction was universal in ESRD. However, few studies clarified the association of T cell dysfunction and clinical outcomes. This study is aim to explore valuable markers of T cell dysfunction predicting bad clinical outcomes including death, cardiovascular disease, infection and tumor. Hopefully, these finding will provide foundation for further mechanism research and better therapeutic options for ESRD patients in the future.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) suffer from high morbidity and mortality of cardiovascular and infectious disease and increased risk of all-cause mortality which is mainly attributed to the disturbed immune response. More and more evident indicated that T cell dysfunction was universal in ESRD. Recent evidence suggests uremia-related immune changes resemble to aging immune system, increasing immunological age of T cells by 20-30 years. As compared to an age-matched healthy control, ESRD patients present a lower thymic output of naïve T cells, a decline in the T-cell telomere length and an increase in the differentiation status towards the terminal differentiated memory phenotype with a large number of CD28-negative T cells. More importantly, these changes are strongly associated with a history of cardiovascular diseases and the occurrence of severe infectious episodes in this population, supporting the idea that T cell dysfunction is a critical feature in this population and will impact clinical outcomes profoundly. This study prospectively researched the predictive value of T cell dysfunction for all-cause mortality and clinical complication in hemodialysis (HD) patients.

ELIGIBILITY:
Inclusion Criteria:

* had been on hemodialysis treatment for at least 6 months in Blood Purification Center,Zhongshan Hospital, Fudan University

Exclusion Criteria:

* underwent any kind of cardiovascular or infection event in three months
* with hematological diseases, rheumatic diseases, active malignancies
* with history of human immunodeficiency virus infection
* currently use of any immunosuppressants
* not followed-up at Zhongshan Hospital, Fudan University

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * aged 18 years and older
  * had been on hemodialysis treatment for at least 6 months in our blood purification center
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | January 2021 to December 2023
  mortality during the study

SECONDARY OUTCOMES:
Cardiovascular disease | January 2021 to December 2023
  having documented congestive heart failure, coronary artery disease, peripheral arterial occlusive disease, or stroke
Infection event | January 2021 to December 2023
  having new onset of infections which requiring standard intravenous antibiotics or hospitalization
Cancer | January 2021 to December 2023
  having new discovered tumors

CONTACTS AND LOCATIONS:
Overall Officials: Bo Shen, MD, Study Director — Fudan University; Fangfang Xiang, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No